CLINICAL TRIAL: NCT03097120
Title: The Estrogen Replacement and Atherosclerosis Trial
Brief Title: The Estrogen Replacement and Atherosclerosis Trial ; Primary Outcome Measure is Mean Minimal Coronary Artery Diameter After Avg of 3.2 Yrs.
Acronym: ERA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U01HL45488
Record Dates: First submitted 2011-04-26; First posted 2017-03-31 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2018-07

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- unopposed estrogen (Active Comparator): 0.625 mg of conjugated equine estrogen
  Interventions: Drug: 0.625 mg of conjugated equine estrogen
- estrogen-plus-medroxyprogesterone (Active Comparator): 0.625 mg of conjugated equine estrogen plus 2.5 mg of medroxyprogesterone acetate
  Interventions: Drug: 0.625 mg of conjugated equine estrogen plus 2.5 mg of medroxyprogesterone acetate
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo tablets

INTERVENTIONS:
Drug: 0.625 mg of conjugated equine estrogen — one tablet containing 0.625 mg of conjugated equine estrogen and a placebo tablet daily
  Arms: unopposed estrogen
Drug: 0.625 mg of conjugated equine estrogen plus 2.5 mg of medroxyprogesterone acetate — one tablet of 0.625 mg of conjugated equine estrogen plus one tablet 2.5 mg of medroxyprogesterone acetate daily
  Arms: estrogen-plus-medroxyprogesterone
Drug: placebo tablets — two placebo tablets daily
  Arms: placebo

SUMMARY:
Background: Heart disease is a major cause of illness and death in women. To understand better the role of estrogen in the treatment and prevention of heart disease, more information is needed about its effects on coronary atherosclerosis and the extent to which concomitant progestin therapy may modify these effects.

Methods: The investigators randomly assigned a total of 309 women with angiographically verified coronary disease to receive 0.625 mg of conjugated estrogen per day, 0.625 mg of conjugated estrogen plus 2.5 mg of medroxyprogesterone acetate per day, or placebo. The women were followed for a mean (±SD) of 3.2±0.6 years. Base-line and follow-up coronary angiograms were were analyzed by quantitative methods. Follow-up coronary angiograms were obtained after an average of 3.2 years of follow up.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal
* not currently receiving estrogen-replacement treatment
* one or more epicardial coronary stenoses of at least 30 percent of the luminal diameter, as measured by quantitative coronary angiography

Exclusion Criteria:

* known or suspected breast or endometrial carcinoma
* previous or planned coronary-artery bypass surgery,
* a history of deep-vein thrombosis or pulmonary embolism,
* symptomatic gallstones,
* serum aspartate aminotransferase level more than 1.5 times the normal value,
* fasting triglyceride level of more than 400 mg per deciliter
* serum creatinine level of more than 2.0 mg per deciliter
* more than 70 percent stenosis of the left main coronary artery,
* uncontrolled hypertension, or
* uncontrolled diabetes.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 1995-01; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
mean minimal coronary-artery diameter | at average of 3.2 years follow-up
  mean minimal coronary-artery diameter within each subject at follow-up, analyzed on an intention-to-treat basis

SECONDARY OUTCOMES:
stenosis as a percentage of the reference diameter | at average of 3.2 years follow-up
development of new lesions in a patient | at average of 3.2 years follow-up
Models focusing on change in diameter were also examined | at average of 3.2 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David M. Herrington, MD, MHS, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Herrington DM, Reboussin DM, Klein KP, Sharp PC, Shumaker SA, Snyder TE, Geisinger KR. The estrogen replacement and atherosclerosis (ERA) study: study design and baseline characteristics of the cohort. Control Clin Trials. 2000 Jun;21(3):257-85. doi: 10.1016/s0197-2456(00)00054-4. PMID 10822123
- [Result] Herrington DM, Reboussin DM, Brosnihan KB, Sharp PC, Shumaker SA, Snyder TE, Furberg CD, Kowalchuk GJ, Stuckey TD, Rogers WJ, Givens DH, Waters D. Effects of estrogen replacement on the progression of coronary-artery atherosclerosis. N Engl J Med. 2000 Aug 24;343(8):522-9. doi: 10.1056/NEJM200008243430801. PMID 10954759